CLINICAL TRIAL: NCT00124228
Title: Effects of Intravenous Albumin Administration on Renal Function and Survival in Patients With Cirrhosis and Infections Unrelated to Spontaneous Bacterial Peritonitis. A Prospective, Stratified, Randomized and Controlled Study.
Brief Title: Albumin Administration in Patients With Cirrhosis and Infections Unrelated to Spontaneous Bacterial Peritonitis
Acronym: Infecir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Fondo Investigación Sanitaria España, 05/0273
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIS05/0273; FIS
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-08

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; Infection; Sepsis; Renal failure
MeSH Terms: conditions — Fibrosis; Infections; Sepsis; Renal Insufficiency | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Antibiotic following hospital Protocols according the cause of the infection .
- 2 (Active Comparator): Antibiotic following hospital Protocols according the cause of infection plus albumin
  Interventions: Drug: Human Albumin

INTERVENTIONS:
Drug: Human Albumin — albumin 1.5g/kg body weight the first day of inclusion plus 1g/kg/body weight the 3th day of inclusion.
  Arms: 2

SUMMARY:
Spontaneous bacterial peritonitis (SBP) present in cirrhotic patients induces severe circulatory dysfunction, which results in renal failure in up to 30% of the patients. Renal failure is an important prognostic marker, representing the major predictive factor of in-hospital mortality.

Recent studies have shown that plasma volume expansion with albumin associated with cefotaxime in patients with SBP is more efficient to prevent renal failure than cefotaxime treatment alone. The in-hospital and three-month mortality rates, furthermore, were significantly lower in the group treated with albumin.

It is not known if other bacterial infections unrelated to SBP represent a risk factor for the development of renal failure among cirrhotic patients. The researcher's group has recently performed a study to evaluate the incidence, characteristics and outcome, of renal failure in patients with cirrhosis and bacterial infections unrelated to SBP associated with the systemic inflammatory response syndrome (Terra, unpublished results). Among a total of 106 patients, 29 (27%) presented renal failure during the course of infection. Renal failure was characterized by intense renal vasoconstriction (intrarenal resistive index of 0.83 +/- 0.09, measured by Doppler ultrasound), reduction of mean arterial pressure and an important activation of endogenous vasoconstriction systems. The three-month survival probability of patients with infection and renal failure was 34 %, much lower than that of patients with infection but not presenting renal failure (87%, p<0.0001). These results suggest that the development of renal failure in patients with cirrhosis and bacterial infections different from SBP, associated with signs of a systemic inflammatory response, is very frequent and results in a very poor prognosis. Taken as a whole, these data strongly indicate the need to consider these patients as candidates for liver transplantation and to plan strategies for its prevention.

The objective of this project, therefore, is to evaluate if the plasma volume expansion with albumin, associated with conventional antibiotic therapy, can prevent the development of renal failure and increase survival rates in cirrhotic patients with bacterial infections unrelated to spontaneous bacterial peritonitis.

DETAILED DESCRIPTION:
Recent studies have shown that the administration of cefotaxime (first choice treatment for SBP) associated with plasma volume expansion with albumin in patients with SBP, was more efficient to prevent renal failure than cefotaxime treatment alone (10% vs. 33%, respectively). The in-hospital and three-month mortality rates, furthermore, were significantly lower in the group treated with albumin (10% vs. 29% and 22% vs. 41%, respectively). There was a significant increase in the plasma renin activity in the group treated with cefotaxime alone as compared to the group receiving cefotaxime associated with the expansion with albumin. A direct relationship between plasma renin activity levels and the development of renal failure was also observed.

Based on the previous information the main objective of this study is to evaluate if the plasma volume expansion with albumin associated to conventional antibiotics therapy, can prevent the development of renal failure and increase survival rates in cirrhotic patients with bacterial infections unrelated to spontaneous bacterial peritonitis. If that proves to be the case, albumin should be administered as first choice treatment associated with antibiotics to all the cirrhotic patients with bacterial infection and systemic inflammatory response syndrome.

Other parameters to be investigated include:

* In-hospital mortality.
* Evaluation of the treatment effects over the renal vascular territory, estimated by Doppler ultrasonography of the intrarenal arteries.
* Evaluation of the relationship between the development of renal failure and the activity of endogenous vasoactive systems: plasma renin activity, plasma concentration of aldosterone, noradrenaline, atrial natriuretic factor and nitrites. Evaluation of the relationship between the development of renal failure and the concentration of inflammatory cytokines: tumor necrosis factor-α, interleukin-6, interleukin-1, interleukin-10.
* Evaluation of heart function and its relationship with the development of renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Cirrhosis defined by clinical, analytical or histological criteria;
* Active infection defined by the presence of at least two of the criteria for systemic inflammatory response syndrome (SIRS), necessarily including neutrophilia in the hemogram. In case of a positive culture, the presence of only one of the SIRS criteria is considered sufficient for the infection diagnosis. SIRS is defined by: temperature >38º or <36º C, heart beat >90 beats/min, breath frequency >20 resp/min, white cell count >12000/mm3 or <4000/mm3 or >6% of immature cells.
* Written informed consent.
* Absence of the exclusion criteria described below

Exclusion Criteria:

* Use of antibiotics during the week preceding the study, except for prophylaxis of spontaneous bacterial peritonitis;
* Hepatocarcinoma: hepatocarcinoma patients presenting more than 3 nodes > 3 cm, or one node larger than 5 cm, tumoral portal thrombosis or extrahepatic tumor extension;
* Heart insufficiency or advanced chronic obstructive pulmonary disease;
* Digestive bleeding during the week preceding the study;
* Presence of septic shock, defined as: sepsis with hypotension (systolic pressure <90 mm Hg or a decrease >40 mm Hg as compared to the basal pressure), in spite of an adequate liquid reposition, signs of a poor peripheral perfusion or need of vasoactive drugs;
* Plasma creatinine > 3 mg/dL;
* Severe dehydration (defined by a central venous pressure < 3 cm H2O due to severe diarrhea or to a strong response to diuretic treatment) at inclusion in the study; the patients with PVC lower than 3 will receive plasma volume expansion with saline and will be reevaluated within 24 h. If the expansion is able to correct PVC (defined as PVC > 3), the patients will be apt to be included in the study.
* Existence of diseases which can influence the short term survival.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Renal failure rate | During hospitalization
  presence of renal failure at admision or development during hospitalization
Renal failure rate | at 3 month
  outcome of renal failure 3 months after inclusion in the study

SECONDARY OUTCOMES:
In-hospital and at 3 month mortality | During hospitalization and 3-month mortality
Evaluation of the treatment effects over the renal vascular territory | at the end of antibiotic treatment (infection resolution)
  Renal resistence index will be determined at baseline and at the end of treatment
Evaluation of the relationship between the development of renal failure and the activity of endogenous vasoactive systems | At baseline, at day 3rd and at the end of treatment
  Evaluation of vasoactive systems and the development or presence of renal failure. These relationships will be evaluated at baseline, at day 3rd and at the end of antibiotic treatment
Evaluation of the relationship between the development of renal failure and the concentration of inflammatory cytokines | At baseline, at day 3rd and at the end of treatment
  Evaluation of cytokines levels and the development or presence of renal failure. These relationships will be evaluated at baseline, at day 3rd and at the end of antibiotic treatment
Evaluation of heart function and its relationship with the development of renal failure | At baseline and at the end of treatment
  Evaluation of heart function and the development or presence of renal failure. These relationships will be evaluated at baseline, and at the end of antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, Dr, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Guevara M, Terra C, Nazar A, Sola E, Fernandez J, Pavesi M, Arroyo V, Gines P. Albumin for bacterial infections other than spontaneous bacterial peritonitis in cirrhosis. A randomized, controlled study. J Hepatol. 2012 Oct;57(4):759-65. doi: 10.1016/j.jhep.2012.06.013. Epub 2012 Jun 23. PMID 22732511